CLINICAL TRIAL: NCT00268684
Title: A Phase III Trial Comparing Whole Brain Radiation (WBRT) and Stereotactic Radiosurgery (SRS) Alone Versus With Temozolomide or Erlotinib in Patients With Non-Small Cell Lung Cancer and 1-3 Brain Metastases
Brief Title: Comparison Study of WBRT and SRS Alone Versus With Temozolomide or Erlotinib in Patients With Brain Metastases of NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Radiation Therapy Oncology Group (Network)
Other Study IDs: TASMC-05-FB-05235-CTIL
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2005-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Erlotinib Hydrochloride; Temozolomide

INTERVENTIONS:
Drug: Erlotinib, Temozolomide

SUMMARY:
The objectives of the study is to determine if either temozolomide or erlotinib combined with WBRT and SRS improves survival as compared to WBRT and SRS alone.Ptients with histologically confirmed NSCLC with the presence of 1-3 intraparenchymal brain metastases will be randomized to 3 arms. All of the patients will receive WBRT and SRS. The patients of the arm 1 will receive radiation treatment only, the arm 2 patients will be treated with temozolomide and arm 3 patients will receive erlotinib

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer with the presence of 1-3 intraparenchymal brain metastases.
2. A contrast-enhanced MRI demonstrating the presence of 1-3 brain metastases performed within two weeks prior to registration.
3. The contrast-enhancing intraparenchymal brain tumor must be well circumscribed and must have a maximum diameter of ≤ 4.0 cm in any direction on the enhanced scan. If multiple lesions are present and one lesion is at the maximum diameter, the other(s) must not exceed 3.0 cm in maximum diameter.
4. Patients who present with symptoms of brain metastases at the time of initial diagnosis are eligible and do not need to demonstrate one month of stable scans.
5. Age 18 years or older.
6. Zubrod 0-1
7. Neurologic Function Status 0, 1, or 2.
8. Patients may have stable extracranial metastases.
9. Contrast-enhancing CT scans of the chest, abdomen and pelvis, and bone scan to determine the extent of extracranial malignant disease.
10. Adequate bone marrow reserve
11. Patients randomized to receive erlotinib who are on enzyme inducing seizure medicines including phenytoin, carbamazepine, rifampicin, barbiturates must be converted to a nonenzyme inducing anti-seizure medication. Patients on Arm 3 will not be able to start treatment immediately if converting.
12. Patient must sign a study-specific informed consent form. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative.

    -

Exclusion Criteria:

1. Major medical illnesses or psychiatric impairment
2. Patients who have undergone a complete resection of all known brain metastases.Patients who have undergone subtotal resection are eligible providing residual disease is =/< 4.0 cm in maximum diameter.
3. Inability to obtain histologic proof of NSCLC.
4. Patients with leptomeningeal metastases documented by MRI or CSF evaluation.
5. Clinical or radiographic evidence of progression (other than the study lesion(s)) within one month prior to enrollment. (Patients who have brain metastases at initial presentation are eligible and do not need to demonstrate one month of stable scans).
6. Patients with metastases within 10 mm of the optic apparatus so that some portion of the optic nerve or chiasm would be included in the high dose SRS boost field.
7. Patients with metastases in the brainstem, midbrain, pons, or medulla.
8. Patients with liver metastases.
9. Previous cranial radiation.
10. Women who are pregnant or nursing
11. Patients who are HIV positive are not eligible.
12. Any evidence of clinically active interstitial lung disease
13. Treatment with a non-approved or investigational drug within 30 days before Day 1 of studytreatment.
14. Concomitant use of St. John's Wort.
15. History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib and temozolomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381
Dates: Start 2005-05

PRIMARY OUTCOMES:
survival

CONTACTS AND LOCATIONS:
Overall Officials: Felix Bokstein, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel